CLINICAL TRIAL: NCT04948398
Title: Post-Trial Access for Guselkumab in Patients With Familial Adenomatous Polyposis Who Are Experiencing Clinical Benefit After Completing 48 Weeks of Treatment in CNTO1959COR1001
Brief Title: Post-Trial Access for Guselkumab in Participants With Familial Adenomatous Polyposis
Status: No longer available | Type: Expanded Access
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108964; CNTO1959APC4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-06-24; First posted 2021-07-02 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Adenomatous Polyposis Coli
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — guselkumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Guselkumab — Guselkumab 100 milligrams (mg) will be administered subcutaneously once every 8 weeks.

SUMMARY:
The purpose of this post-trial access (PTA) program is to provide guselkumab to participants with Familial Adenomatous Polyposis (FAP) who are experiencing clinical benefit after completing 48 weeks of treatment in Study CNTO1959COR1001.

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC